CLINICAL TRIAL: NCT01225068
Title: An Exploratory Randomized Placebo Controlled Trial of Milnacipran in Patients With Chronic Neuropathic Low Back Pain
Brief Title: Effect of Milnacipran in Chronic Neuropathic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Forest Laboratories (Industry); Shirley Ryan AbilityLab (Other); Best Practice (Unknown)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00036897
Record Dates: First submitted 2010-10-13; First posted 2010-10-20 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran (Experimental): milnacipran 50 mg bid; can be increased to 100 mg bid
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Total of 100 mg (50 mg twice a day) for 6 weeks. Option to increase to 200 mg (100 mg twice a day) after two weeks of treatment. Includes gradual escalation and discontinuation for week 1 and after week 6.
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — 2 matching pills per day for 6 weeks. Option to increase dose after two weeks of treatment. Includes gradual escalation and discontinuation for week 1 and after week 6.
  Arms: Placebo

SUMMARY:
Low back pain is a public health problem affecting between 70-85% of adults at some time in their life. This study is being done to study the safety and effectiveness of the drug Milnacipran in treating chronic low back pain.

DETAILED DESCRIPTION:
This exploratory study aims to evaluate Milnacipran in individuals with chronic neuropathic low back pain. A sample of 40 individuals with chronic low back pain will be enrolled in a double-blind, randomized, parallel group study comparing twice daily administration of milnacipran with placebo (total 100 mg bid-or equivalent placebo dosing). The study will last 6 weeks with subjects being evaluated at the start of the study, at the end of a one-week drug-free period, and at 1, 2 and 6 weeks of treatment. Additionally, subjects will evaluated after treatment has ended. Both standard endpoint outcome measures as well as validated daily self-report measures of pain and activity/disability will be utilized.

ELIGIBILITY:
Inclusion Criteria:

1. History of low back pain for a minimum of 6 months with radiation to leg or buttocks
2. Over 18 years of age and under 70
3. Must have a visual analogue scale (VAS) pain score >50mm
4. Must be in generally stable health
5. Must be willing to abstain from alcohol during the course of the study
6. If female, must be post-menopausal, or practicing a highly effective method of contraception or abstinence during the course of the study
7. Must be able to read and understand instructions and the questionnaires
8. Must be willing to participate in daily data collection requirements via telephone (IVRS)
9. Must understand all aspects of the study, and willing to sign an informed consent form in that regard.

Exclusion Criteria:

1. Low back pain associated with systemic signs or symptoms (e.g. fever or chills)
2. Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, history of surgery or tumor in the back
3. Involvement in litigation regarding back pain or other disability claim, or receiving workmen's compensation, or seeking either as a result of low back pain.
4. Neurological disorder including history of seizures
5. Major psychiatric disorder during the past six months
6. Active suicidal ideation or recent suicidal behavior
7. Significant other medical disease such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease or malignancy
8. Significant renal disease or severe renal insufficiency
9. History of, or current, substance abuse/dependence
10. Significantly abnormal laboratory values
11. Pregnant or lactating any time during the course of the study
12. Known sensitivity to Savella or other SNRI
13. Glaucoma
14. Taking any MAOI, sibutramine, digoxin, tricyclic antidepressants, other SNRI, Opioids.
15. Beck Depression Inventory Score >30
16. Current Sleep Disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient clinic
Pre-assignment Details: Screening visit prior to randomization
Groups:
- Milnacipran: Milnacipran : Total of 100 mg (50 mg twice a day) for 6 weeks. Option to increase to 200 mg (100 mg twice a day) after two weeks of treatment. Includes gradual escalation and discontinuation for week 1 and after week 6.
- Placebo: Placebo treatment group
Period: Overall Study
Arm/Group | Milnacipran | Placebo
Started | 20 | 20
Completed | 16 | 19
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.6) | 48.3 (9.1) | 47.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Effect Size of VAS Pain
Description: Effect size (ES) calculation for VAS pain between milnacipran and placebo groups' ES is dimensionless; Visual analogue scale (VAS) measured pain in integral units from 0 (low end) to 100 (high end); ES (Cohen's d) is a well described statistical construct and is calculated from the difference between the means (determined at baseline and 6 weeks here) divided by the pooled standard deviation.
  This is the primary outcome measure.
Time Frame: 6 weeks from baseline
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 19 | 16
units on a scale | 24.8 (32.5) | 31.3 (26.4)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; effect size is endpoint and not comparison; Test type: Superiority or Other; effect size is endpoint and not comparis — no p value for effect size calculations ES is dimensionless; ES (Cohen's d) is a well described statistical construct and is calculated from the difference between the means (here at baseline and 6 weeks) divided by the pooled standard deviation; no p value for effect size calculations; effect size = 0.22

ADVERSE EVENTS:
Time Frame: baseline to 8 weeks after randomization
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 14/20 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=20) | Placebo (N=20)
colon resection (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=20) | Placebo (N=20)
headache (General disorders) | 2 (2) | 7 (7)
nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 3 (3)
constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
drowsiness (General disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No